CLINICAL TRIAL: NCT02811458
Title: A Pragmatic Randomized Controlled Trial of Group Transdiagnostic Cognitive-Behavior Therapy for Anxiety Disorders in Primary Care
Brief Title: Clinical Trial of Transdiagnostic Cognitive-Behavior Therapy for Anxiety Disorders
Acronym: T-CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Estrie University Integrated Health and Social Services Center - University Hospital of Sherbrooke (Other); CISSS de Laval (Unknown); Integrated University Health and Social Services Center of the Capitale-Nationale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIHR-340410; CIHR-334091 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2016-05-24; First posted 2016-06-23 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Panic Disorder; Agoraphobia; Social Anxiety Disorder; Generalized Anxiety Disorder
Keywords: Panic Disorder; Agoraphobia; Social Anxiety Disorder; Generalized Anxiety Disorder; Cognitive-Behavioral Therapy
MeSH Terms: conditions — Panic Disorder; Agoraphobia; Phobia, Social; Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transdiagnostic CBT (Experimental): Group psychotherapy according to the Transdiagnostic Cognitive-Behavioral Therapy treatment protocol (Norton, 2012)
  Interventions: Behavioral: Transdiagnostic Cognitive-Behavioral Therapy
- Treatment-as-usual (No Intervention): Treatment-as-usual and a differed intervention (if desired by participants) after the 8-month follow up.

INTERVENTIONS:
Behavioral: Transdiagnostic Cognitive-Behavioral Therapy — Treatment in the Transdiagnostic CBT condition will consist of 12 weekly 2-hour sessions following the manualized treatment protocol including psychoeducation, cognitive restructuring, exposure and relapse prevention.
  Arms: Transdiagnostic CBT

SUMMARY:
Anxiety disorders are the most common mental disorders in community settings, and they are associated with significant psychological distress, functional and social impairment. Although pharmacological and psychological treatments for anxiety and depression have existed for several years now, only a minority of anxiety disorder sufferers are treated according to guidelines. Cognitive behavior therapy (CBT) is the most consistently efficacious psychological treatment for anxiety disorders, but implementation of CBT in primary care is challenging due to limited resources. Recent studies indicate that transdiagnostic group CBT for multiple anxiety disorders could be a promising alternative to individual CBT in primary care. The aim of the study is to examine the effectiveness of group CBT for anxiety disorders as a complement to usual care. The clinical trial will be conducted in three Health and Social Services Centers in the province of Québec (i.e. Sherbrooke, Laval and Québec). Patients will be French-speaking adults with anxiety disorders, and they will be randomly assigned to one of two treatment conditions: a) Transdiagnostic group CBT (12 weekly 2-hour sessions), b) usual care. The transdiagnostic group CBT will be offered as a differed intervention to participants in the usual care group after the 8-month follow up. Participants in both study arms will undergo a baseline clinical evaluation as well as outcome assessment interviews at post-treatment, 4, 8, and 12 month follow-up time-points. The primary study results will include improvement on a questionnaire on anxiety symptoms. Widespread implementation of group CBT could lead to better outcomes for a large number of patients living with anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 (upper age limit added 2016-11-18)
* Fluent in spoken and written French.
* Meeting DSM-5 diagnostic criteria for at least one of the following anxiety disorders as a primary mental disorder: Panic Disorder, Agoraphobia, Generalized Anxiety Disorder and/or Social Anxiety Disorder according to a clinical rating ≥ 4 for the Anxiety Disorders Interview Schedule for DSM-5 (ADIS-5) administered by a trained PhD-level clinician.

Exclusion Criteria:

* Active suicidal intentions, psychosis, bipolar disorder, active substance-related disorder and addictive disorder in the past 12 months (sections or screening questions in ADIS-5).
* Marked cognitive impairment [Épreuve des 5 mots (Dubois, 2002) administered in case of doubt by assessor].
* Consultation with a psychiatrist in the past 12 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Change in Beck Anxiety Inventory (BAI) | Baseline and post-treatment; within two weeks after the 12th treatment session, based on the timeframe of the intervention group (treatment completion)
Change in Clinical Severity Rating from the Anxiety Disorders Interview Schedule for DSM-5 - Adult Version (ADIS-5) | Baseline and post-treatment; within two weeks after the 12th treatment session, based on the timeframe of the intervention group (treatment completion) (Outcome 2 added 2017-12-12)

SECONDARY OUTCOMES:
Change in Beck Anxiety Inventory (BAI) | Baseline, post-treatment, 4-month, 8-month and 12-month follow-ups
Change in Clinical Severity Rating from the Anxiety Disorders Interview Schedule for DSM-5 - Adult Version (ADIS-5) | Baseline, post-treatment and 8-month follow-ups
Change in Panic Disorder Severity Scale (Self-Report) | Baseline, post-treatment, 4-month, 8-month and 12-month follow-ups
Change in Mobility Inventory for Agoraphobia | Baseline, post-treatment, 4-month, 8-month and 12-month follow-ups
Change in Penn State Worry Questionnaire | Baseline, post-treatment, 4-month, 8-month and 12-month follow-ups
Change in Social Phobia Inventory | Baseline, post-treatment, 4-month, 8-month and 12-month follow-ups
Change in Patient Health Questionnaire (PHQ-9) | Baseline, post-treatment, 4-month, 8-month and 12-month follow-ups
Change in EuroQol (EQ-5D-5L) | Baseline, post-treatment, 4-month, 8-month and 12-month follow-ups
Change in Administrative databases records | Starting 12 months prior to participant enrollment up to the 12-month follow-up
  Beneficiary registry (sex, birthdate, and death registry), Med-Écho hospitalizations (diagnosis, procedures), medical services (physician, diagnosis, acts, services) and pharmaceutical services (medication, dose, duration).
Change in Anxiety Disorder Diagnostic Questionnaire - weekly version (ADDQ-W) | ADDQ-W administered weekly over the course of the 12 weekly group therapy sessions to assess change in anxiety severity.

CONTACTS AND LOCATIONS:
Overall Officials: Pasquale Roberge, Ph.D., Principal Investigator — Université de Sherbrooke; Martin D. Provencher, Ph.D., Principal Investigator — Laval University
Locations (3):
- Canada (3):
  - Centre intégré de santé et de services sociaux de Laval, Laval, Quebec
  - Centre intégré universitaire de santé et de services sociaux de l'Estrie, Sherbrooke, Quebec
  - Centre intégré universitaire de santé et de services sociaux de la Capitale-Nationale, Québec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roberge P, Provencher MD, Gosselin P, Vasiliadis HM, Gaboury I, Benoit A, Antony MM, Chaillet N, Houle J, Hudon C, Norton PJ. A pragmatic randomized controlled trial of group transdiagnostic cognitive-behaviour therapy for anxiety disorders in primary care: study protocol. BMC Psychiatry. 2018 Oct 3;18(1):320. doi: 10.1186/s12888-018-1898-1. PMID 30285672
- [Derived] Chapdelaine A, Vasiliadis HM, Provencher MD, Norton PJ, Roberge P. Moderators of the cost-effectiveness of transdiagnostic CBT for anxiety disorders over an 8-month time horizon using a net-benefit regression framework. BMC Health Serv Res. 2023 Jun 8;23(1):596. doi: 10.1186/s12913-023-09468-7. PMID 37291599
- See also: BMC Psychiatry — https://bmcpsychiatry.biomedcentral.com/articles/10.1186/s12888-018-1898-1